CLINICAL TRIAL: NCT00417391
Title: Phase II Study of RR110 in Patients With Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R&R Inc. (Industry)
Responsible Party: Miwako Ishido/Manager, R&R Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1101-01
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — N2,N6-bis(4-(2-aminoethoxy)quinolin-2-yl)-4-((4-fluorobenzyl)oxy)pyridine-2,6-dicarboxamide; tamibarotene

ARMS (2):
- 1 mg RR110 (Experimental): 1 mg RR110
  Interventions: Drug: RR110 (Tamibarotene)
- 4 mg RR110 (Experimental): 4 mg RR110
  Interventions: Drug: RR110 (Tamibarotene)

INTERVENTIONS:
Drug: RR110 (Tamibarotene) — 1 mg RR110
  Other Names: Tamibarotene; Am80
  Arms: 1 mg RR110
Drug: RR110 (Tamibarotene) — 4 mg RR110
  Other Names: Tamibarotene; Am80
  Arms: 4 mg RR110

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and pharmacokinetics profile of 1 and 4 mg/kg/day RR110 administrated orally for 8 weeks in patients with active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CDAI score ranging from 220 to 450
* Patients with CRP > 1 mg/dL
* Patients who can be hospitalized at least 2 weeks after first administration

Exclusion Criteria:

* Patients who have previously used anti-TNF antibody, cyclosporine, methotrexate or tacrolimus within 12 weeks of screening
* Patients who have had surgical bowel resections within 4 weeks of screening
* Patients who have previously used total parental nutrition or more than 900 kcal/day of enteral nutrition within 4 weeks of screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change in Crohn's disease active index (CDAI) score | 8 weeks

SECONDARY OUTCOMES:
Rate of clinical response as defined by CDAI decrease > 70 or 100 from baseline | 8 weeks
Rate of clinical remission as defined by CDAI < 150 | 8 weeks
Change in CRP, SAA, and fibrinogen levels, and IBDQ and CDEIS scores | 10 weeks
Safety parameters | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshifumi Hibi, M.D., Ph.D., Study Chair — Keio University
Locations (8):
- Japan (8):
  - Toyohashi, Aichi-ken
  - Sakura, Chiba
  - Sapporo, Hokkaido
  - Nishinomiya, Hyōgo
  - Fujisawa, Kanagawa
  - Nakagami, Okinawa
  - Ōtsu, Shiga
  - Shinjuku, Tokyo